CLINICAL TRIAL: NCT06197919
Title: Effects of Posture Exercises With and Without Breathing Exercises in Forward Head Posture
Brief Title: Effect of Posture and Breathing Exercises in Forward Head Posture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/23/0169
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Forward Head Posture
Keywords: breathing exercises
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: participants of both group are informed about possible risk and potential benefits but don't know which group they are placed in. assessors are also masked. concealment will be done via sealed opaque method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postural exercises with breathing exercises (Experimental): The postural exercise program consisted of two strengthening and stretching exercises. The exercises involved chin tucks in, shoulder retraction , and unilateral and bilateral pectoralis stretches alternating each 2-week period. 36 Participants were instructed to complete 3 sets of 12 repetitions of the strengthening exercises and 3 stretching exercises held for 30 seconds each.
  For the breathing exercises in experimental group, breathing program includes respiratory muscle training, relaxation techniques, breathing techniques, e.g., deep breathing, hand controlled abdominal/diaphragmatic breathing, aimed stretching and strengthening exercises are combined with each other. Deep breathing, controlled diaphragmatic breathing, slow relaxed exhalation with pursed lips technique, direct apnoea exercises and segmental breathing techniques. exercise protocol will be continued for 10 weeks with and initial, after 5 weeks and final assessment of pain and CVA.
  Interventions: Other: postural exercises with breathing exercises
- postural exercises without breathing exercises (Experimental): In this study forward head posture will be defined as CVA<49°, which was diagnosed by photogrammetry method.
  The postural exercise program consisted of two strengthening and stretching exercises. The exercises involved
  (a) chin tucks in (c) shoulder retraction , and (d) unilateral and bilateral pectoralis stretches alternating each 2-week period. 36 Participants were instructed to complete 3 sets of 12 repetitions of the strengthening exercises and 3 stretching exercises held for 30 seconds each. This program was to be repeated 4 times per week. They also returned for a consultation every 2 weeks to be checked for exercise technique and progression, if appropriate. Progress to the next exercise level was indicated if the participant could complete 12 repetitions, 3 times easily with correct form.
  Interventions: Other: postural exercises

INTERVENTIONS:
Other: postural exercises — In this study forward head posture will be defined as CVA<49°, which was diagnosed by photogrammetry method.
  The postural exercise program consisted of two strengthening (deep cervical flexors and shoulder retractors) and two stretching (cervical extensors and pectoral muscles) exercises based on Kendall et al's approach. The exercises involved
  1. chin tucks ins
  2. a chin drop in sitting
  3. shoulder retraction
  4. unilateral and bilateral pectoralis stretches Participants were instructed to complete 3 sets of 12 repetitions of the strengthening exercises and 3 stretching exercises held for 30 seconds each. This program was to be repeated 4 times per week. They also returned for a consultation every 2 weeks to be checked for exercise technique and progression, if appropriate. Progress to the next exercise level was indicated if the participant could complete 12 repetitions, 3 times easily with correct form
  Arms: postural exercises without breathing exercises
Other: postural exercises with breathing exercises — The postural exercise program consisted the exercises i.e chin tucks in, a chin drop in sitting, shoulder retraction. Participants were instructed to complete 3sets of 12repetitions of these exercises. This program was to be repeated 4times per week. They also returned for a consultation every 2weeks to be checked for exercise technique and progression, if appropriate. Progress to the next exercise level was indicated if the participant could complete 12repetitions, 3times easily with correct form.
  For the breathing exercises in experimental group, breathing program includes respiratory muscle training, relaxation techniques, breathing techniques, e.g., deep breathing, hand controlled diaphragmatic breathing, relaxation technique, deep breathing, controlled diaphragmatic breathing, slow relaxed exhalation with pursed lips technique, and segmental breathing techniques. exercise protocol will be continued for 6 weeks with and initial, after 3weeks and final assessment of pain and CVA.
  Arms: postural exercises with breathing exercises

SUMMARY:
This study aims to compare the effects of postural exercises with and without breathing exercises in the subjects having forward head posture.

DETAILED DESCRIPTION:
Forward head posture (FHP) is a prevalent postural deviation that can occur in individuals of various age groups, spanning from childhood to old age. It manifests as an anterior positioning of the head in relation to the neck in the sagittal plane. . FHP is commonly associated with the excessive extension of the upper cervical spine (C1-C3) and flexion of the lower cervical spine (C4-C7). A common method to diagnose forward head posture is by measuring craniovertebral angle i.e. if CVA<49 than FHP is positive. In many cases faulty postures are linked with different musculoskeletal conditions as well as breathing difficulties. Forward head posture specifically impairs the mobility and functionality of the diaphragm, resulting in inefficient contraction of abdominal muscles and reduced lung capacity. A randomized clinical trial will be conducted so that we can rule out proper treatment protocol for forward head posture.

For this randomized clinical trial, 36 participants having forward head posture will be recruited from Sehat medical complex and shalamar hospitals Lahore by nonprobability convenient sampling. Participants will divide in two groups A and B by randomization. Group A will be given both exercise regimes of postural exercises and breathing exercises while group B will be given with only postural exercise protocol. Pain, ROM and craniovertebral angle will be assessment before the treatment start, after 5 weeks and at the end of treatment after 10 weeks. After the collection of data in 8 months, Statistical analysis using SPSS version 21, will be done to summarize the results.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with 20 to 35 years of age, both male and female
* Individuals with CVA <49.

Exclusion Criteria:

* History of Surgery of thorax or spine or both.
* Traumatic neck injury.
* Acute or chronic neuro-muscular pain.
* Clinical deformity present in thoracic cage or spine

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
photogrammetry for CVA and cervical range of motion(ROM) (image j) | 6 weeks
  CVA, can be measured using the lateral photo exposing C7 and the ear. The participants will maintain the natural head posture through the measurement method of self balance posture.It is the angle made by the line that connects the seventh cervical spine with the tragus and the horizontal line of 7th cervical spine in the standing position. A CVA is of ,49 is characterized as Forward head posture.
  image j is an image processing and analysis program that can read both image file formats and raw formats. it has been introduces as a reliable assessment tool used to measure cervical angle in several studies on forward head posture.

SECONDARY OUTCOMES:
Numeric pain rating scale (NPRS): | 6 weeks
  The NPRS is a subjective pain rating scale using an 11 point scale from 0 to 10, where 0 means "no pain" and 10 means "intolerable pain". Participants select the whole number that best represent their level of pain. The reliability is>0.95 with ICC value 0.86-0.95
Goniometer | 6 weeks
  Goniometer is an objective tool to measure range of motion of different joints of body. it has good reliability (r = .70)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza, MS, Principal Investigator — Riphah International University; izzah ijaz, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Sehat Medical Complex, Lahore, Punjab Province
  - Shalamar Hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No